CLINICAL TRIAL: NCT02036372
Title: PILGRIM - Perioperative Insulin, GIK or GLP-1 Treatment in Diabetes Mellitus Type II
Brief Title: Perioperative Insulin, GIK or GLP-1 Treatment in Diabetes Mellitus
Acronym: PILGRIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, B Preckel, Prof dr B Preckel, MD, PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL 41467.018.12
Record Dates: First submitted 2014-01-10; First posted 2014-01-15 (Estimated); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Diabetes Mellitus Type II
Keywords: glucose; diabetes mellitus; perioperative
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Liraglutide; Insulin Aspart; Glucose; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- BR (bolus regimen) (Experimental): * Day before surgery: half evening dose long acting insulin
  * Day of surgery:
    * patients using mealtime and longacting insulin/NPH: withhold mealtime morning dose, stop glucose lowering tablets
    * patients using only long acting insulin/NPH: half dose of long-acting or NPH insulin, stop glucose lowering tablets
  * Measure blood glucose every 60 minutes, start 30 min prior to surgery
  * Give bolus of insulin according to treatment algorithm
  Interventions: Drug: Insulin bolus
- LG (Liraglutide) (Experimental): * Day before surgery: half dose of long acting and mealtime insulin from start liraglutide
  * Day of surgery: withhold own insulin, stop oral glucose lowering tablets
  * Start with 0.6 mg liraglutide subcutaneously (s.c.) the day prior to surgery at 17.00hr.
  * In case of nausea graded higher than minimal, the patient will be excluded from the study
  * Otherwise, treatment will be continued with 1.2 mg liraglutide s.c. per day on the day of surgery at 07.00hr.
  * Measure glucose every 60 minutes, start 30 min prior to surgery
  * Adjust according to bolus algorithm of BR group
  Interventions: Drug: Liraglutide; Drug: Insulin bolus
- GIK (glucose -insulin - potassium) infusion (Active Comparator): * Day before surgery: half evening dose long acting insulin
  * Day of surgery: stop oral glucose lowering tablets and withhold own insulin.
  * GIK infusion: 500 cc glucose 5% with insulin and 10 mmol KCL per 500 cc. Start at 83 ml/hr.
  * Calculate the insulin amount in the GIK infusion according to the formula:
  I= (PG-7)/(200/W)+8 I=Insulin amount, PG=glucose 30 minutes preoperative, W= body weight in kg
  * Measure blood glucose every 60 minutes, start 30 min prior to surgery
  * Adjust glucose > 8 mmol/l according to treatment algorithm
  Interventions: Drug: GIK infusion

INTERVENTIONS:
Drug: Liraglutide
  Other Names: Victoza
  Arms: LG (Liraglutide)
Drug: Insulin bolus
  Other Names: novorapid
  Arms: BR (bolus regimen); LG (Liraglutide)
Drug: GIK infusion — continuous infusion
  Other Names: glucose, insulin, potassium infusion
  Arms: GIK (glucose -insulin - potassium) infusion

SUMMARY:
The incidence of diabetes mellitus type II is increasing. More and more patients who need surgery have diabetes mellitus type II. Despite an enormous amount of glucose lowering protocols and the proven negative effects of hyperglycaemia. There is no evidence for the optimal glucose lowering protocol.

This study investigates the optimal intraoperative treatment algorithm to lower glucose in patients with diabetes mellitus type 2 undergoing non-cardiac surgery, comparing intraoperative glucose-insulin-potassium infusion (GIK), insulin bolus regimen (BR) and GLP-1 (liraglutide, LG) treatment.

DETAILED DESCRIPTION:
Diabetes mellitus is associated with poor outcome after surgery. The prevalence of diabetes in hospitalised patients is up to 40%, meaning that the anaesthesiologist will encounter a diabetes patient in the operating room on a daily basis. Multiple protocols for perioperative glucose regulation have been developed, ranging from intravenous glucose-insulin-potassium infusion to subcutaneous bolus regimens. Despite this abundance of published glucose lowering protocols and the proven negative effects of intraoperative hyperglycaemia in diabetes, there is no evidence regarding the optimal intraoperative glucose lowering treatment. Recently, incretins have been introduced to lower blood glucose. The main hormone of the incretin system is glucagon-like peptide-1 (GLP-1). GLP-1 increases insulin and decreases glucagon secretion in a glucose-dependent manner, resulting in low incidence of hypoglycaemia. This study investigates for the first time the optimal intraoperative treatment algorithm to lower glucose in patients with diabetes mellitus undergoing non-cardiac surgery.

Objective:

This study investigates the optimal intraoperative treatment algorithm to lower glucose in patients with diabetes mellitus type 2 undergoing non-cardiac surgery, comparing intraoperative glucose-insulin-potassium infusion (GIK), insulin bolus regimen (BR) and GLP-1 (liraglutide, LG) treatment.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* known diabetes mellitus type II for > 3 months
* aged 18-75 years
* scheduled for elective non-cardiac surgery

Exclusion Criteria:

- Daily insulin dosage of > 1 IU/kg body weight

* Oral corticosteroid use
* Planned for day-care (ambulant) surgery
* Planned ICU stay post-operatively
* Planned bowel surgery
* History of chronic pancreatitis or idiopathic acute pancreatitis
* Impaired renal function defined as serum-creatinine ≥ 133 μmol/L for males and ≥ 115 μmol/L for females
* Females of child bearing potential who are pregnant, breast-feeding or intend to become pregnant or are not using adequate contraceptive methods (adequate contraceptive measures as required by local law or practice)
* Known or suspected allergy to trial product(s) or related products
* Any condition that the local investigator feels would interfere with trial participation or the evaluation of results

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Median glucose | 1 hour after surgery
  The difference in median glucose between the GIK + BR and LG group 1 hour after surgery

SECONDARY OUTCOMES:
Total Insulin administration | 1 day postoperative
  The difference in insulin administration between the GIK + BR and LG group within 24 h after start of surgery
Median glucose | 4 hours and 1 day postoperative
  The difference in median glucose between the GIK + BR and LG group 4 hours and 1 day after surgery
Postoperative complications | 1 month after surgery
  The difference in proportion of any postoperative complication within the first month
Hypoglycemia | From start treatment until the morning of day 1 postoperative
  The occurrence of mild and severe hypoglycemia (glucose <4.0 mmol/l and <2.3 mmol/l, respectively) during and up to 24 h after surgery
Hypo- and hyperkalemia | from start treatment until morning of day 1 postoperative
  The occurrence of hypokalemia (<3.5 mmol/l) and hyperkalemia (>5.0 mmol/l) during and up to 24 h after surgery
Glucose | From start treatment until morning of day 1 postoperative
  the difference in median glucose 1hr preoperative, 1, 4 hours postoperative, 1 day postoperative between the three groups.

CONTACTS AND LOCATIONS:
Overall Officials: Benedikt Preckel, MD, PhD, Principal Investigator — Academic Medical Centre - AMC-UvA
Locations (3):
- Netherlands (3):
  - Academic Medical Center Amsterdam, Amsterdam, Please Select
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Diakonessenhuis, Utrecht

REFERENCES:
- [Derived] Polderman JA, Houweling PL, Hollmann MW, DeVries JH, Preckel B, Hermanides J. Study protocol of a randomised controlled trial comparing perioperative intravenous insulin, GIK or GLP-1 treatment in diabetes-PILGRIM trial. BMC Anesthesiol. 2014 Oct 14;14:91. doi: 10.1186/1471-2253-14-91. eCollection 2014. PMID 25419179
- See also: American Diabetes Association — https://diabetes.org/